CLINICAL TRIAL: NCT02042482
Title: The Effect of the Nutritional Supplements: Ultra Q10 and L-carnitine on the Clinical Course of Myelodysplastic Syndrome
Brief Title: The Effect of Combination Ultra Q10 and L-carnitine on the Course of Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Dr Kalman Filanovsky, MD, Kaplan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMC01-35-12
Record Dates: First submitted 2014-01-15; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Myelodysplastic Syndrome
Keywords: Ultra coenzyme Q10; L-carnitine
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coenzyme Q10U, L-carnitine (Experimental): Patients receive combination of coenzyme Q10U 180 milligram and L-carnitine 2000 milligram
  Interventions: Dietary Supplement: Coenzyme Q10U, L-carnitine

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10U, L-carnitine

SUMMARY:
The purpose of this study is determine whether combination Q10 , L-carnitine and multivitamin and mineral complex is effective in treatment of patients with low and intermidiate1-2 risk Myelodysplastic syndrome

DETAILED DESCRIPTION:
The primary objectives of this study are to assess response (as measured by increase in blood counts, cytogenetic/molecular changes in the bone marrow, improved endurance) to the supplements treatment.

The secondary objectives are to determine:

Quality of life assessment(FACT: QOL Questionnaire) Cancer fatigue reduction. Physiological functioning assessment Rate and depth transfusion reduction Duration of response. Time to progression. Overall survival. Estimated cytokine profile and another immunological and biochemical parameters of mitochondrial function before and after six months of treatment.

ELIGIBILITY:
Inclusion Criteria:

Patient willing and able complies with the protocol requirements. Patient given voluntary written informed consent before performance of any study-related procedure that is not part of standard medical care; with the understanding that the consent may be withdrawn by the patient at any time without prejudice to their future medical care.

Patient is older than 18 years at the time of signing the informed consent. Patients older than 80 years will sign informed consent after psycho-geriatric evaluation.

Patient diagnosed with Myelodysplastic syndrome, Low risk and intermediate-1risk according to international prognostic scoring system with hemoglobin level less than 11g/l or platelets less than 100000/ mcl or absolute neutrophils count less than 1000/mcl. With or without fatigue syndrome.

INT-2 and high risk patients may be included into this trial when they are not eligible for other treatment except Best Supportive Cure or failure to other conventional treatment approach.

Bone marrow aspiration examination including cytogenetics performed up to 12 months before inclusion and absence clinic-laboratory evidence of progressive disease in last month Patient has a life-expectancy > 3 months

Exclusion Criteria:

Any serious medical conditions, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he or she participates in this study or confounds the experimental ability to interpret data from the study.

Pregnant or lactating females. Prior history of malignancies, other than MDS, unless the subject has been free of the disease for ≥ 3 years. Exceptions include the following: Basal cell carcinoma of the skin, Squamous cell carcinoma of the skin, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histological finding of prostate cancer (TNM stage of T1a or T1b).

Bone marrow blast count >30%. Patient has known active infectious hepatitis B or C, or HIV infection Administration of investigational drugs in the last 3 months. High risk MDS patients and INT-2 patients who are candidates for cytoreductive or epigenetics treatment.

Any psychological, sociological condutions likely to affect compliance with the study follow-up schedule.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Hemoglobin, Platlets,White blood counts | 12 weeks,24 weeks

SECONDARY OUTCOMES:
Overall response rate | 24 weeks
Progression free survival | 24 weeks,52 weeks
Duration of response | 24 weeks 52 weeks
Quality of life. | 12 weeks 24 weeks 36weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kalman Kalman, MD, Principal Investigator — Kaplan Medical Center, Institute of hematology
Locations (1):
- Kaplan Medical Center, Rehovot, Israel